CLINICAL TRIAL: NCT02643472
Title: GPS (Giving Parents Support): Parent Navigation After NICU Discharge
Acronym: GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Fratantoni, MD, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IHS-1403-11567
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-02

CONDITIONS: Premature Birth of Newborn; Family; Immature Newborn; Newborn Morbidity; Infant Newborn Disease
Keywords: neonate; newborn; neonatal intensive care unit; NICU; NICU discharge; parent navigator; peer to peer; peer coaching
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Notebook (Other): Parents of infants who were discharged from the Children's National NICU will be randomized to receive enhanced usual care by provision of a NICU care resource notebook. Parents will be notified about group assignment prior to discharge. Stratification will occur according to birth weight.
  Interventions: Behavioral: Care Notebook
- Care Notebook + Parent Navigator (Experimental): Parents of infants who were discharged from the Children's National NICU will be randomized to receive a care notebook + Parent Navigation. Parents will be notified about group assignment prior to discharge. Stratification will occur according to the birth weight.
  Interventions: Behavioral: Parent Navigator; Behavioral: Care Notebook

INTERVENTIONS:
Behavioral: Parent Navigator — Parents will be contacted by the parent navigator within 2 business days after discharge to assess how the family is coping, answer questions, and provide necessary resources. Navigators will be in touch with families monthly and according to the parent's needs. They will assist the parent in making and keeping appointments, answer questions about insurance coverage, medical equipment and supplies, and serve as a liaison between parent and healthcare providers. However, the specific PN intervention for each family will be based on each family's needs and therefore may differ.
  Other Names: Peer to Peer Support
  Arms: Care Notebook + Parent Navigator
Behavioral: Care Notebook — A care notebook will be provided to all parents at discharge. The notebook was created to provide resources and serve as an organizer for appointments for parents of NICU graduates. It was based on peer to peer feedback from former NICU parents, in addition, to community resources developed by current Parent Navigator Program at Children's National Health System.

SUMMARY:
BACKGROUND: Annually >400,000 US newborns require neonatal intensive care unit (NICU) care.1/3 will require ongoing or specialty care after discharge. Some NICU graduates can be classified as children with special health care needs (CSHCN) who will require health and related services of a type or amount beyond that required by children generally. NICU parents report increased anxiety and stress during their stay and transition home from the NICU. Short-term peer-to -peer programs during hospitalization decrease stress, anxiety and depression for mothers, however, no studies have evaluated the effects of long term post-discharge peer support. Children's National (CN) provides medical home services to CSHCN through its Parent Navigator Program (PNP). Parent Navigators (PNs) are CSHCN parents who provide peer emotional support, access to community resources, and assistance with navigating complicated health systems. NICU graduates and their caregivers may benefit from support provided by PNs after discharge. No data regarding the impact of PNs on patient and family outcomes of the NICU graduate are available.

OBJECTIVE: To assess the impact of a PNP on a parent's self-efficacy, stress, anxiety, depression; infant health care utilization, and immunization status.

METHODS: 300 NICU graduates will be randomized to receive either PN for 12 months (intervention group) or usual care (comparison group). Baseline data at 1 week, 1, 3, 6, and 12 months after discharge will be collected from caregivers in both groups including scales for self-efficacy, stress, anxiety, and depression, infant healthcare utilization and immunization status. Outcomes will be compared at 12 months.

PATIENT OUTCOMES (PROJECTED) The study outcomes are parental self-efficacy, stress, anxiety, and depression; infant health care utilization and immunization status.

ANTICIPATED IMPACT Prior studies utilizing small samples have suggested that peer support in the NICU can reduce anxiety and depression in caregivers. It is unclear whether peer support after discharge, when a family is faced with the total care of their child without structured supports, can significantly impact parents' ability to care for their child. The investigators anticipate that this simple intervention will increase self-efficacy in caregivers, reduce stress, anxiety, and depression, in turn resulting in improved health outcomes for their child.

DETAILED DESCRIPTION:
Specific Aims:

Infants who are discharged from the neonatal intensive care unit (NICU) almost invariably have high levels of health care needs in the first year after discharge, requiring multiple sub specialist visits, medications, and/or medical technology needs. Parents of NICU infants are often overwhelmed by the needs of their infants after they are discharged home and frequently have few supports to help them cope. This study will investigate the impact of peer to peer support through a Parent Navigation program for NICU graduates and their parents. The study aims will be achieved through a randomized controlled trial of Parent Navigation using a care resource notebook as the control intervention.

The specific aims of this study are to:

1. Determine if Parent Navigation increases overall parental self-efficacy and decreases stress among parents caring for a child with a special health care need (CSHCN) when measured at repeated time points during the 12 months after NICU discharge.

   Hypothesis 1a: Parent Navigation will increase parental self-efficacy, when compared with the control group.

   Hypothesis 1b: Parent Navigation will decrease parenting stress, when compared with the control group.
2. Determine if Parent Navigation improves overall levels of anxiety and depression in parents of children with special health care needs when measured repeatedly during the 12 months after NICU discharge.

   Hypothesis 2a: Parent Navigation will improve parent anxiety, compared with control group.

   Hypothesis 2b: Parent Navigation will lessen parent depression, compared with control group.
3. Determine if Parent Navigation positively impacts on infant health outcomes during the 12 months after NICU discharge.

Hypothesis 3a: Parent Navigation/Intervention group will have significantly fewer hospitalizations when compared with control group.

Hypothesis 3b: Parent Navigation will have significantly fewer emergency department (ED) visits, when compared with control group.

Hypothesis 3c: Parent Navigation will result in improved immunization status, when compared with control group.

Hypothesis 3d. By supporting parents' emotional function, infant developmental progress will be enhanced.

Background :

NICU parents experience high levels of stress, anxiety, and depression, and low levels of self-efficacy. Neonates comprise one of the largest groups of medically complex infants in the United States. Of the 4 million live births in 2012, 11.5% (~460,000) were born preterm at < 37 weeks gestation. The District of Columbia alone has a higher rate (12.8%) of preterm infants, which is 11% higher than the national average. The vast majority of infants born preterm and ~1% of full term infants with significant illnesses at birth (e.g., congenital anomalies) will require care in a neonatal intensive care unit (NICU), and ~30% of infants being discharged from the NICU ("NICU graduates") annually (110,000 babies) require supplementary short -term or ongoing specialty care and have increased risk of long- term disability, including cerebral palsy, deafness, blindness, and neurodevelopmental impairment. At discharge, this large cohort of neonates and their families face tremendous challenges as they transition from a highly structured medical environment to a less structured home environment. Some challenges identified include feeling unprepared to care for their infant at home despite extensive teaching in the NICU setting, feeling socially isolated as the typical celebratory process of giving birth and going home with baby has been disrupted by a serious medical condition and prolonged hospital stay. Additionally, depression and anxiety among mothers of infants have been shown to be associated with infant feeding difficulties, suboptimal parenting practices, and altered health care utilization.

Parent navigation is a unique patient -centered intervention in which parents with experience caring for their own child with special health care need offer peer to peer support and mentoring to another parent of a child with a special health care need. In 2008, Children's National instituted a Parent Navigation program, in which Parent Navigators (PNs), who are parents of children with special health care needs, are employed by CN to provide peer to peer support to other parents of children with special health care need . These parents provide their own personal experience and expertise in navigating the often confusing and frustrating health care systems. Although the PN model is based on self-efficacy and social support models, there are no published studies on the impact of PN on parental self-efficacy, depression, stress, and infant health outcomes. The investigators believe that neonates and their caregivers would benefit from peer to peer support provided by PNs after discharge. Currently, there are no data regarding the impact of PNs on patient and family outcomes of the NICU graduate.

Preliminary Studies:

As a first phase of this study, the investigators conducted focus groups with parents of recently discharged NICU infants (4 focus groups, n=18 participants), parent navigators (1 focus group n=3), parents (n=2), NICU social workers, case managers, and nurses (1 focus group, n=23); NICU providers (1 focus group, n=5) and community providers (n=2). The investigators' intervention is informed by this data.

ELIGIBILITY:
Inclusion Criteria:

* parents of neonates receiving care in the Children's National NICU

Exclusion Criteria:

* infant is not being discharged with a custodial parent (e.g., in custody of Child Protection Services)
* neither parent can complete an interview in English,
* the parent who will be providing most of the care is younger than 18 years of age,
* those with insufficient knowledge of English to participate in the telephone interviews
* the parent/caregiver has plans to leave the District of Columbia (DC) metropolitan area permanently within the following year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fratantoni, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Younge T, Jacobs M, Tuchman L, Streisand R, Soghier L, Fratantoni K. Sociodemographic risk factors, parental stress and social support in the neonatal intensive care unit. Arch Dis Child Fetal Neonatal Ed. 2023 Mar;108(2):165-169. doi: 10.1136/archdischild-2022-324119. Epub 2022 Sep 6. PMID 36805477
- [Derived] Fratantoni K, Soghier L, Kritikos K, Jacangelo J, Herrera N, Tuchman L, Glass P, Streisand R, Jacobs M. Giving parents support: a randomized trial of peer support for parents after NICU discharge. J Perinatol. 2022 Jun;42(6):730-737. doi: 10.1038/s41372-022-01341-5. Epub 2022 Mar 8. PMID 35260824
- [Derived] Carty CL, Soghier LM, Kritikos KI, Tuchman LK, Jiggetts M, Glass P, Streisand R, Fratantoni KR. The Giving Parents Support Study: A randomized clinical trial of a parent navigator intervention to improve outcomes after neonatal intensive care unit discharge. Contemp Clin Trials. 2018 Jul;70:117-134. doi: 10.1016/j.cct.2018.05.004. Epub 2018 May 5. PMID 29733982

RESULTS

PARTICIPANT FLOW:
Groups:
- Care Notebook: Parents of infants who were discharged from the Children's National NICU will be randomized to receive enhanced usual care by provision of a NICU care resource notebook. Parents will be notified about group assignment prior to discharge. Stratification will occur according to birth weight.
  Care Notebook: A care notebook will be provided to all parents at discharge. The notebook was created to provide resources and serve as an organizer for appointments for parents of NICU graduates.
- Care Notebook + Parent Navigator: Parents of infants who were discharged from the Children's National NICU will be randomized to receive a care notebook + Parent Navigation (PN). Parents will be notified about group assignment prior to discharge. Stratification will occur according to the birth weight.
  Parent Navigator: Parents will be contacted by the parent navigator within 2 business days after discharge to assess how the family is coping, answer questions, and provide necessary resources. Navigators will be in touch with families monthly and according to the parent's needs. The specific PN intervention for each family will be based on each family's needs and therefore may differ.
  Care Notebook: A care notebook will be provided to all parents at discharge. The notebook was created to provide resources and serve as an organizer for appointments for parents of NICU graduates.
Period: Overall Study
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Started | 150 | 150
Completed | 123 | 116 (One participant completed CESD-10 but not other measures at 12 months; n=115 for other measures.)
Not Completed | 27 | 34
Not completed — Death | 2 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 22 | 26

BASELINE CHARACTERISTICS:
Groups:
- Care Notebook + Parent Navigator: Parents of infants who were discharged from the Children's National NICU will be randomized to receive a care notebook + Parent Navigation. Parents will be notified about group assignment prior to discharge. Stratification will occur according to the birth weight.
  Parent Navigator: Parents will be contacted by the parent navigator within 2 business days after discharge to assess how the family is coping, answer questions, and provide necessary resources. Navigators will be in touch with families monthly and according to the parent's needs. The specific PN intervention for each family will be based on each family's needs and therefore may differ.
  Care Notebook: A care notebook will be provided to all parents at discharge. The notebook was created to provide resources and serve as an organizer for appointments for parents of NICU graduates.
- Total: Total of all reporting groups
Arm/Group | Care Notebook | Care Notebook + Parent Navigator | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent age
  years | 30.4 (6.5) | 29.9 (6.5) | 30.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Parent sex
  Participants
    Female | 129 | 138 | 267
    Male | 21 | 12 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Parent race
  Participants
    Race: American Indian/Pacific Islander | 6 | 2 | 8
    Race: Asian | 11 | 6 | 17
    Race: Black | 66 | 67 | 133
    Race: White | 56 | 61 | 117
    Race: Mixed race/not reported | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300
Education [Count of Participants; unit: Participants] — Parent education
  Participants
    High school or less | 34 | 43 | 77
    Trade/vocational/some college | 46 | 41 | 87
    College degree or more | 70 | 66 | 136
Relationship [Count of Participants; unit: Participants] — Parent relationship
  Participants
    Single | 22 | 27 | 49
    Married/partnered | 128 | 123 | 251
Other children [Count of Participants; unit: Participants] — Presence of other children in parent household
  Participants
    No other children at home | 68 | 61 | 129
    At least one other child | 82 | 89 | 171
Infant gestational age [Count of Participants; unit: Participants]
  <32 weeks | 39 | 33 | 72
  32-36 weeks | 23 | 36 | 59
  >=37 weeks | 88 | 81 | 169
Infant birth weight [Count of Participants; unit: Participants]
  <1500 grams | 32 | 31 | 63
  1500-2499 grams | 34 | 29 | 63
  >=2500 grams | 84 | 90 | 174
Infant sex [Count of Participants; unit: Participants]
  Male | 88 | 86 | 174
  Female | 62 | 64 | 126
Infant length of stay category [Count of Participants; unit: Participants]
  <=1 week | 40 | 38 | 78
  8-17 days | 32 | 41 | 73
  18-47 days | 38 | 37 | 75
  >=48 days | 40 | 34 | 74

OUTCOME MEASURES:

1. Primary Outcome: Parental Self-Efficacy
Description: Parental self-efficacy was measured using the Perceived Maternal Parenting Self-Efficacy Questionnaire (PMPS-E). Mean scores were determined and compared between groups. PMPS-E scores can range from 20-80, and higher scores indicate higher levels of parental self-efficacy.
Time Frame: baseline; 1 week, 1 month, 3 months, 6 months, 12 months after discharge
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Care Notebook + Parent Navigator: Parents of infants who were discharged from the Children's National NICU will be randomized to receive a care notebook + Parent Navigation. Parents will be notified about group assignment prior to discharge. Stratification will occur according to the birth weight.
  Parent Navigator: Parents will be contacted by the parent navigator within 2 business days after discharge to assess how the family is coping, answer questions, and provide necessary resources. Navigators will be in touch with families monthly and according to the parent's needs. They will assist the parent in making and keeping appointments, answer questions about insurance coverage, medical equipment and supplies, and serve as a liaison between parent and healthcare providers. However, the specific PN intervention for each family will be based on each family's needs and therefore may differ.
  Care Notebook: A care notebook will be provided to all parents at discharge. The notebook was created to provide resources and
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 123 | 115
score on a scale
  Predicted means: main effect of group | 74.94 [74.20 to 75.68] | 74.75 [73.96 to 75.55]
  Estimated scores: 1-week | 72.7 [71.9 to 73.6] | 72.6 [71.7 to 73.5]
  Estimated scores: 1-month | 73.8 [73.0 to 74.6] | 73.6 [72.8 to 74.5]
  Estimated scores: 3-month | 76.0 [75.3 to 76.8] | 75.9 [75.1 to 76.7]
  Estimated scores: 6-month | 78.0 [77.3 to 78.8] | 77.9 [77.1 to 78.7]
  Estimated scores: 12-month | 76.9 [76.1 to 77.6] | 76.7 [75.9 to 77.6]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.73, Generalized Estimating Equations; In analyzing predicted means, results of Generalized Estimating Equations (GEE) modeling controlled for time from baseline at each assessment

2. Secondary Outcome: Parental Anxiety
Description: Parental anxiety was measured using the State Trait Anxiety Inventory (STAI). Mean scores were determined and compared between groups. The trait portion (Y-2) was only administered at baseline, while the state portion (Y-1) was administered at every interval and used for longitudinal analyses. STAI scores can range from 20-80, and higher scores indicate higher levels of anxiety.
Time Frame: baseline; 1 week, 1 month, 3 months, 6 months, 12 months after discharge
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 123 | 115
score on a scale
  Predicted means: main effect of group | 29.55 [28.24 to 30.87] | 31.14 [29.68 to 32.61]
  Estimated scores: 1-week | 31.0 [29.6 to 32.3] | 32.5 [31.0 to 34.0]
  Estimated scores: 1-month | 30.2 [28.9 to 31.6] | 31.8 [30.3 to 33.2]
  Estimated scores: 3-month | 28.7 [27.3 to 30.1] | 30.2 [28.6 to 31.8]
  Estimated scores: 6-month | 27.4 [25.9 to 29.0] | 28.9 [27.2 to 30.7]
  Estimated scores: 12-month | 28.7 [27.0 to 30.4] | 30.2 [28.5 to 32.0]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; STAI Y-1 data was used in these statistical analyses; Test type: Superiority; p = 0.12, Generalized Estimating Equations; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Parental Stress
Description: Parental stress was measured using the Parental Stress Scale (PSS). Mean scores were determined and compared between groups. PSS scores can range from 18-90, and higher scores indicate higher levels of parental stress.
Time Frame: baseline; 1 week, 1 month, 3 months, 6 months, 12 months after discharge
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 123 | 115
score on a scale
  Predicted means: main effect of group | 27.47 [26.34 to 28.60] | 29.29 [28.16 to 30.42]
  Estimated scores: 1-week | 28.6 [27.4 to 29.7] | 30.4 [29.2 to 31.5]
  Estimated scores: 1-month | 28.0 [26.8 to 29.1] | 29.8 [28.6 to 30.9]
  Estimated scores: 3-month | 26.7 [25.5 to 27.9] | 28.5 [27.3 to 29.7]
  Estimated scores: 6-month | 25.7 [24.5 to 27.0] | 27.5 [26.3 to 28.8]
  Estimated scores: 12-month | 27.1 [25.8 to 28.4] | 28.9 [27.5 to 30.2]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.03, Generalized Estimating Equations; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: General Stress
Description: General stress was measured using the Perceived Stress Scale (PSS-10), a 10-item instrument which asks respondents to consider their feelings and thoughts during the last month. Total scores range from 0-40, with higher scores indicating higher levels of stress
Time Frame: baseline, 1 week, 1 mo, 3 mo, 6 mo, 12 months after discharge
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 123 | 115
score on a scale
  Predicted means: main effect of group | 12.51 [11.56 to 13.46] | 13.74 [12.78 to 14.70]
  Estimated scores: 1-week | 14.3 [13.3 to 15.3] | 15.5 [14.5 to 16.4]
  Estimated scores: 1-month | 13.3 [12.4 to 14.3] | 14.5 [13.5 to 15.4]
  Estimated scores: 3-month | 11.2 [10.2 to 12.3] | 12.4 [11.3 to 13.4]
  Estimated scores: 6-month | 9.6 [8.5 to 10.8] | 10.8 [9.6 to 11.9]
  Estimated scores: 12-month | 11.9 [10.7 to 13.1] | 13.0 [11.8 to 14.2]

5. Secondary Outcome: Parental Stress in the Neonatal Intensive Care Unit
Description: The Parental Stressor Scale:Neonatal Intensive Care Unit (PSS:NICU) was used to measure NICU-specific stress. Mean total and subscale scores were determined using Metric 1 (applicable stress) and compared between groups. PSS:NICU scores can range from 1-5, and higher scores indicate higher levels of NICU-specific stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 148 | 148
score on a scale | 2.11 (0.92) | 1.99 (0.80)

6. Secondary Outcome: Parental Depression
Description: Parental depression was measured using the 10-item Center for Epidemiological Study Depression Scale (CES-D 10). Mean scores were determined and compared between groups. CES-D 10 scores can range from 0-30, and a score >=10 indicates the presence of depressive symptoms.
Time Frame: baseline; 1 month, 3 months, 6 months, 12 months after discharge
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 123 | 116
score on a scale
  Predicted means: main effect of group | 6.04 [5.34 to 6.73] | 6.98 [6.29 to 7.68]
  Estimated scores: 1-month | 6.9 [6.2 to 7.6] | 7.8 [7.1 to 8.5]
  Estimated scores: 3-month | 5.3 [4.6 to 6.0] | 6.2 [5.4 to 6.9]
  Estimated scores: 6-month | 4.0 [3.3 to 4.8] | 5.0 [4.1 to 5.8]
  Estimated scores: 12-month | 6.2 [5.3 to 7.1] | 7.1 [6.2 to 8.0]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.06, Generalized Estimating Equations; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: ED Visits
Description: Infant ED visits were parent-reported and totaled over a period of 12 months.
Time Frame: One year
Measure: Median (Inter-Quartile Range); unit: ED visits
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 147 | 145
ED visits | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Hospitalizations
Description: Infant hospitalizations were parent-reported and totaled over a period of 12 months.
Time Frame: One year
Measure: Median (Inter-Quartile Range); unit: Hospitalizations
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 147 | 145
Hospitalizations | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Infant Immunization Status
Description: Infant immunization status was either provider-reported or accessed via a state registry. The number of neonates with a complete immunization series within 12 months after discharge were compared between groups. Complete immunization status was defined as receipt of 3 diphtheria tetanus acellular pertussis (DTaP) vaccines, 3 pneumococcal conjugate vaccines (PCV13), and either 2 or 3 Hemophilus influenzae b (HIB) vaccines, depending on vaccine type (e.g. PedvaxHIB at 2 and 4 months, ActHIB at 2, 4, and 6 months).
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 143 | 136
Participants
  Fully immunized | 107 | 98
  Not fully immunized | 36 | 38
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Test type: Superiority; p = 0.60, Chi-squared

10. Secondary Outcome: Infant Developmental Status
Description: Infant developmental status was measured using the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley III). The Bayley III was administered between 11-13 months of study follow-up, and it used corrected infant age to account for prematurity. Composite scores for cognitive, language, and motor domains were determined and compared between groups. Bayley scores can range from 40-160, and higher scores indicate higher levels of infant development.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
Number analyzed (Participants) | 65 | 62
score on a scale
  Cognitive | 97.83 (16.25) | 98.13 (17.13)
  Language | 88.49 (15.33) | 86.89 (17.49)
  Motor | 91.26 (16.02) | 91.79 (18.98)
Statistical Analysis 1: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Infant development status was evaluated with Bayley subscales. Cognitive subscale; Test type: Superiority; p = 0.92, t-test, 2 sided
Statistical Analysis 2: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Infant development status was evaluated with Bayley subscales. Language subscale; Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 3: Comparison: Care Notebook vs Care Notebook + Parent Navigator; Infant development status was evaluated with Bayley subscales. Motor subscale; Test type: Superiority; p = 0.87, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period of 12 months.
Description: The deaths of these infants were unrelated to our study. This study was minimal risk, offering peer support after NICU discharge, and did not involve any medical procedures or interventions.
Arm/Group | Care Notebook | Care Notebook + Parent Navigator
All-Cause Mortality (participants affected / at risk) | 2/150 | 5/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02643472/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02643472/SAP_001.pdf